CLINICAL TRIAL: NCT00058357
Title: The Efficacy Of Lidocaine Patch In The Management Of Postsurgical Neuropathic Pain In Patients With Cancer: A Phase III Double-Blind, Crossover Study
Brief Title: Lidocaine Patch in Treating Cancer Patients With Neuropathic Pain After Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NCCTG-N01CB; NCCTG-N01CB; CDR0000288824 (Registry Identifier: NCI Physician Reference Desk)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine patch (Active Comparator): Participants will be instructed to apply a patch or patches (up to 3 maximum simultaneously) directly to the affected area. The patch(es) should be applied during awake hours and then left on continuously for approximately 18 hours or until usual bedtime sleep.
  Interventions: Drug: lidocaine
- Placebo patch (Placebo Comparator): Participants will be instructed to apply a patch or patches (up to 3 maximum simultaneously) directly to the affected area. The patch(es) should be applied during awake hours and then left on continuously for approximately 18 hours or until usual bedtime sleep.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: lidocaine
  Arms: Lidocaine patch
Other: placebo
  Arms: Placebo patch

SUMMARY:
RATIONALE: A lidocaine patch may be effective in relieving numbness, tingling, and other symptoms of neuropathy. It is not yet known whether a lidocaine patch is effective in treating neuropathy in patients who have undergone surgery for cancer.

PURPOSE: This randomized phase III trial is studying lidocaine patch to see how well it works compared to a placebo patch in relieving numbness, tingling, and other symptoms of neuropathy in patients who have undergone surgery for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether a lidocaine patch vs placebo improves postsurgical neuropathic pain in cancer patients.
* Compare the toxic effects of these regimens in these patients.
* Compare the effect of these regimens on mood states, functional abilities, and overall quality of life of these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to etiology of pain (breast surgery vs lung surgery vs amputation vs other), duration of pain (1-3 months vs 4-6 months vs more than 6 months), and current analgesic regimen (opioids [including tramadol] vs antidepressants vs anticonvulsants vs combination vs other vs none). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive a lidocaine transdermal patch (up to 3 patches) applied directly to the painful area for 18 hours once daily. Treatment continues for 4 weeks in the absence of unacceptable toxicity. At the end of week 4, patients cross over to arm II.
* Arm II: Patients receive a placebo transdermal patch applied to the painful area as in arm I. At the end of week 4, patients cross over to arm I.

Pain and quality of life are assessed at baseline and weeks 4 and 8.

Patients are followed at 3-7 days.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Underwent surgical procedure for cancer diagnosis or treatment
* Experiencing persistent pain for at least 1 month

  * Pain must have neuropathic features (e.g., burning, shooting, stabbing, tingling, or pain from light touch)
  * Anatomically related to the surgical site and compatible with nerve injury
  * Pain rating of at least 4 out of 10 on the pain scale
* No pain of multiple etiologies at the proposed treatment site (e.g., pain of neuropathic and muscular or skeletal origin)
* Painful area must be no larger than can be covered by 3 lidocaine patches* NOTE: *Each patch size is 5.5 x 4 inches
* No skin disease, breakdown, infection, or extreme thinning at the site of pain
* No skin or soft tissue malignancy in the painful area

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* At least 6 months

Hematopoietic

* Not specified

Hepatic

* AST ≤ 2 times upper limit of normal

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to understand and complete questionnaires
* No recent history of or concurrent drug or alcohol abuse
* No mental or psychiatric condition that would preclude giving informed consent
* No history of allergic reaction or intolerance to lidocaine or other amide local anesthetics (e.g., bupivacaine)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior neurotoxic chemotherapy* with pain in the same area as postsurgical neuropathic pain, except for pain that was present before neurotoxic chemotherapy administration
* No concurrent neurotoxic chemotherapy* NOTE: *Including taxanes (e.g., paclitaxel or docetaxel), platinum-based compounds (e.g., cisplatin or carboplatin), or vinca alkaloids (e.g., vincristine or vinblastine)

Endocrine therapy

* More than 7 days since prior topical corticosteroids to the painful area
* No new corticosteroids may be initiated during study participation

Radiotherapy

* No concurrent radiotherapy to the painful area

Surgery

* See Disease Characteristics

Other

* More than 7 days since other prior topical medications to the painful area (including capsaicin)
* No change in current analgesic regimen within the past 10 days
* No new analgesic or adjuvant drugs (e.g., antidepressants, anticonvulsants, or anxiolytics) may be initiated during study participation

  * Concurrent stable doses of nonopioid, opioid, and adjuvant analgesic drugs are allowed (including antidepressants or anticonvulsants)
* No concurrent class I antiarrhythmic drugs (e.g., tocainide and mexiletine)
* Concurrent skin lubricants and sunscreen are allowed provided they are not heavily applied

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-05; Primary Completion 2006-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pain intensity rating (NRS) | 4 and 8 weeks

SECONDARY OUTCOMES:
Pain as assessed by the Brief Pain Inventory-Short Form, Neuropathy Pain Scale, Subject Global Impression of Change, Pain Catastrophizing Scale, Profile of Mood States Short Form, and NCCTG Quality of Life | 8 weeks
Incidence of each toxicity reported in each treatment period | 8 weeks
Maximum severity reported of each toxicity | 8 weeks
Distribution of the overall toxicity score | 8 weeks
Proportion of patients who report a preference for lidocaine patch or placebo at study completion | 8 weeks
Proportion of patients who terminate treatment prematurely | up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, MD, Study Chair — Mayo Clinic
Locations (159):
- United States (159):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Providence Hospital, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, P.A. - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, P.A. - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, P.A. - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, P.A. - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, P.A. - Salina, Salina, Kansas
  - Cancer Center of Kansas, P.A. - Wellington, Wellington, Kansas
  - Associates in Womens Health, P.A. - North Review, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Alexandria, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine Associates of Bozeman, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Toledo Surgical Specialists, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - United States Air Force Medical Center Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Cheville AL, Sloan JA, Northfelt DW, Jillella AP, Wong GY, Bearden Iii JD, Liu H, Schaefer PL, Marchello BT, Christensen BJ, Loprinzi CL. Use of a lidocaine patch in the management of postsurgical neuropathic pain in patients with cancer: a phase III double-blind crossover study (N01CB). Support Care Cancer. 2009 Apr;17(4):451-60. doi: 10.1007/s00520-008-0542-x. Epub 2009 Jan 13. PMID 19142669